CLINICAL TRIAL: NCT05716165
Title: Effect of Proprioceptive Knee Braces on the Performance and Endurance of Recreational Soccer Players Aged 60-80 Years
Acronym: FOOTEX60-80
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02522-41
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: knee brace; soccer; aged; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a prospective, monocentric, randomized clinical investigation (order of tests with and without knee braces), carried out in open, over a period of 2 weeks (cohort 1) or 12 weeks (cohort 2), in a population of people aged 60 to 80 years practicing recreational soccer.
Masking Description: the clinical trial is carried out in open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- self-comparison (Experimental): Volunteers will be asked to wear a knee brace on each limb during one of the training sessions. At the end of this training session, a questionnaire will be given to the volunteer to evaluate knee stability, range of motion, confidence when walking, and fear of falling.
  The volunteers will then have to participate in 2 test sessions: one with and one without knee braces.
  The patient will perform tests (Unipodal balance on flat ground, 30s chair stand test, 2,5m up and go test, 6 min-walk) with and without the proprioceptive knee brace in a randomized order.
  At the end of the tests with and without knee brace, a questionnaire will be given to the volunteer to evaluate the stability of the knee, the range of motion, the confidence when walking, the fear of falling, as well as a satisfaction questionnaire about the device.
  There is also a satisfaction questionnaire regarding the proprioceptive knee brace to be completed at the end of the study.
  Interventions: Device: proprioceptive knee braces; Device: No knee brace

INTERVENTIONS:
Device: proprioceptive knee braces — The patient will perform the tests with the knee braces.
Device: No knee brace — The patient will perform the tests without the knee brace.

SUMMARY:
The objective of the study is to evaluate the effect of wearing bilateral proprioceptive knee braces on the endurance of subjects aged 60 to 80 years.

DETAILED DESCRIPTION:
Sporting activity has proven health benefits, particularly for older adults, whose balance and neuromuscular functions decline with age.

On the other hand, physical activity in the elderly population may be hampered by inadequate physical condition, muscle or proprioceptive deficits, or fear of falling or injuring. A proprioceptive knee brace could therefore make physical activity safer and thus improve performance, balance, and ultimately the quality of life of the participants.

The objective of the study is to evaluate the effect of wearing bilateral proprioceptive knee braces on the endurance of subjects aged 60 to 80 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject practicing recreational soccer
* Subject included in the LIBM (inter-university laboratory of motor biology) study: "Effect of recreational soccer practice in persons aged 60 to 80 years"
* Patient whose knee measurements are compatible with the knee brace sizes
* Patient who has signed a free and informed consent form
* Patient affiliated or entitled to a social security plan

Exclusion Criteria:

* Patients with any of the contraindications to the use of the knee brace, as indicated in the instructions for use
* Patient with a major cognitive impairment incompatible with participation in a clinical trial
* Patient participating in another clinical investigation conducted to establish the conformity of a device impacting the judgment criteria
* Vulnerable patient according to article L1121-6 of the public health code, person subject to a legal protection measure or unable to consent freely

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of bilateral proprioceptive knee braces on the endurance of subjects compared to without knee brace. | week 1
  The evaluation of the subjects' endurance corresponds to the difference in results obtained during the 6-minutes walk test in the absence and presence of knee braces.

SECONDARY OUTCOMES:
Evaluate the impact of knee braces on balance compared to without knee brace. | week 1
  Balance will be evaluated via 2 tests:
  * An unipodal balance test performed on flat ground, eyes open and eyes closed, and the result of the test compared in the absence and presence of knee braces.
  * A bipodal test to objectively measure balance, performed on a force platform with eyes open and eyes closed, to determine the projection of the subject's centre of pressure for 30 seconds. The results of the test will be compared in the absence and presence of knee pads.
Evaluate the impact of knee braces on lower limb strength compared to without knee brace. | week 1
  The strength of the lower limbs will be evaluated via the 30s chair stand test and the result of the test compared in the absence and presence of knee braces.
Evaluate the impact of knee braces on walking speed compared to without knee brace. | week 1
  Walking speed and agility will be evaluated during the 2.5m up and go test and the test result compared in the absence and presence of knee braces.
Evaluate the impact of knee braces on the volunteer's feelings about the stability of his knees, their range of motion, his confidence when walking and his fear of falling after the tests and after the training | week 1, week 2
  The feeling of the volunteer will be evaluated via a questionnaire on the stability of the knee, the amplitude of movement, the confidence during the walk and the fear of falling felt after the tests and after the training
Evaluate the influence of the functional capacity of the knees of each volunteer at inclusion on the various performance parameters measured | Day 0
  The functional capacity of the knees at inclusion will be assessed via the Lysholm questionnaire
Evaluate the satisfaction of the volunteers with the device | Last visit
  The volunteers' satisfaction with the system will be evaluated via a specific satisfaction questionnaire.
Evaluate the tolerance of the knee braces | week 1, week 2
  Tolerance will be evaluated through the collection of adverse events following the wearing of knee braces

CONTACTS AND LOCATIONS:
Overall Officials: Roger OULLION, MD, Principal Investigator — Saint-Etienne Jean Monnet University
Locations (1):
- Saint-Etienne Jean Monnet University, Saint-Etienne, France

REFERENCES:
- [Background] Baltaci G, Aktas G, Camci E, Oksuz S, Yildiz S, Kalaycioglu T. The effect of prophylactic knee bracing on performance: balance, proprioception, coordination, and muscular power. Knee Surg Sports Traumatol Arthrosc. 2011 Oct;19(10):1722-8. doi: 10.1007/s00167-011-1491-3. Epub 2011 Apr 6. PMID 21468615
- [Background] Bean JF, Vora A, Frontera WR. Benefits of exercise for community-dwelling older adults. Arch Phys Med Rehabil. 2004 Jul;85(7 Suppl 3):S31-42; quiz S43-4. doi: 10.1016/j.apmr.2004.03.010. PMID 15221722
- [Background] Buchner DM, Cress ME, de Lateur BJ, Esselman PC, Margherita AJ, Price R, Wagner EH. The effect of strength and endurance training on gait, balance, fall risk, and health services use in community-living older adults. J Gerontol A Biol Sci Med Sci. 1997 Jul;52(4):M218-24. doi: 10.1093/gerona/52a.4.m218. PMID 9224433
- [Background] Osoba MY, Rao AK, Agrawal SK, Lalwani AK. Balance and gait in the elderly: A contemporary review. Laryngoscope Investig Otolaryngol. 2019 Feb 4;4(1):143-153. doi: 10.1002/lio2.252. eCollection 2019 Feb. PMID 30828632